CLINICAL TRIAL: NCT06680596
Title: A ctDNA Screening Program in Patients With HR+, HER2 Low Metastatic Breast Cancer for Detection of High-risk Relapse Patients on Any CDK4/6 Inhibitor Followed by a Single Arm Phase II Trial of Trastuzumab-deruxtecan in Patients With Persistent ctDNA After 1 Month of Treatment With Endocrine Therapy Combined With CDK4/6 Inhibitor
Brief Title: Detecting Tumor DNA in the Blood of HR+/HER2-low Metastatic Breast Cancer Patients to Find Candidates for T-DXd Therapy
Acronym: SAFIR3LibHERty
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: AstraZeneca (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GMP-2402; 2024-515349-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Metastatic; Breast Cancer Stage IV
Keywords: HR+; HER2 low; HER2 ultralow; molecular screening; ctDNA; T-DXd; Antibody-drug conjugate; trastuzumab deruxtecan; Breast cancer metastatic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: After an initial screening phase to identify patients with blood circulating tumours persistent, patients will be enrolled in the treatment phase that was designed as an open-label, multicentre, phase II study, to test the efficacy of trastuzumab deruxtecan in terms of progression-free survival (PFS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-DXd (Experimental): T-DXd will be administrated as an intra-venous injection of 5.4 mg/kg every three weeks (1 cycle = 21-day treatment).
  Interventions: Drug: trastuzumab derxutecan

INTERVENTIONS:
Drug: trastuzumab derxutecan — T-DXd will be administrated as an intra-venous injection of 5.4 mg/kg every three weeks (1 cycle = 21-day treatment).

SUMMARY:
After an initial screening phase to identify patients with persistent blood circulating DNA tumors, patients will be enrolled in the treatment phase that was designed as an open-label, multicentre, phase II study, to test the efficacy of trastuzumab deruxtecan in terms of progression-free survival (PFS).

DETAILED DESCRIPTION:
Eligible patients to the screening phase are patients with hormone receptor positive (estrogen receptor and/or progesterone receptor >10%) and HER2 low or ultralow metastatic breast cancer who will receive standard first line therapy with CDK4-6i (any from the market), combined with aromatase inhibitor or fulvestrant. Patient persistence of tumor DNA in the blood at 4 weeks of this standard therapy will be included in the treatment phase with trastuzumab deruxtecan (T-DXd).

ELIGIBILITY:
SCREENING PHASE_________________________________________________________

Inclusion criteria

1. Patient must have signed the written informed consent for screening phase prior to any trial specific procedures.

   Note: When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Patient is ≥18 years of age.
3. Documented breast cancer that:

   * Is metastatic and eligible to biopsy for subsequent histological or cytological confirmation,
   * Is HER2 low (HER2 1+, or 2+ and in situ hybridization (ISH) negative) or HER2 ultra low (IHC 0 with incomplete and faint membrane staining in >0 and ≤10% of tumor cells) on the most recent tumor material available, as defined by the local pathologist under ASCO/CAP guidelines,
   * Is HR-positive (positive for estrogen receptor or progesterone receptor ≥10% of tumor cell nuclei are immunoreactive) in the metastatic setting.
4. Patient has either:

   * a metastatic relapse during or within 1 year after termination of the adjuvant endocrine therapy (AI resistant), or
   * a metastatic relapse more than one year of completing adjuvant AI or a de-novo metastatic breast cancer (AI sensitive/naive).
5. For AI resistant population: patient has previously gone through the ctDNA screening part of the SAFIR 03 - SCREENING/ARRIBA study and fulfilled all the inclusion criteria and none of the exclusion criteria.
6. Patient did not receive any therapy in the metastatic setting.
7. Patient is eligible for a first-line treatment with a marketed CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) in combination with either AI or fulvestrant, according to its marketing authorisation.
8. Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
9. Patient has an adequate bone marrow and organ function.
10. Patient has a measurable or an evaluable disease according to Response Evaluation Criteria In Solid Tumours version 1.1 (RECIST v1.1).
11. Availability of an archived metastatic tumor sample (FFPE) for exploratory research. Bone metastasis are accepted if tissue is representative of tumor tissue (at least 10% tumor cellularity).
12. Patient must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.
13. Registration in a National Health Care System (or equivalent).

Exclusion criteria:

1. Patient is eligible to chemotherapy because of visceral crisis.
2. Patient has a breast cancer amenable for resection or radiation therapy with curative intent.
3. Prior exposure to antibody-drug conjugate or CDK4/6 inhibitors (in metastatic setting). CDK4/6 inhibitors given in adjuvant setting must be stopped for at least 12 months prior screening
4. Patient who has initiated the CDK4/6 inhibitor treatment.
5. Patient is unable to swallow tablets.
6. Patient has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis requiring steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at baseline
7. Patient has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
8. Patient has a history of severe hypersensitivity reactions to other monoclonal antibodies.
9. Person deprived of their liberty or under protective custody or guardianship.
10. Social, familial, or geographic factors that would interfere with study participation or follow-up.

TREATMENT PHASE_________________________________________________________

Inclusion criteria

1. Patient must have signed the written informed consent for the treatment phase prior to any trial specific procedures.

   Note: When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Patient must have discontinued CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) at least 7 days before enrolment, but no longer than 14 days
3. Patients must present a no drop of ctDNA determined by a ctDNA assay after 4 weeks of standard of care treatment with a CDK4/6 inhibitor
4. Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
5. Left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to enrolment.
6. Participant has adequate bone marrow and organ function within 14 days before enrolment, defined as the following laboratory values:

   * Absolute neutrophil count (ANC) ≥1500/mm³,
   * platelet count ≥100,000/mm³,
   * haemoglobin ≥9.0 g/dl,
   * Serum creatinine ≤1.5 × upper limit of normal (ULN) or creatinine clearance ≥30 mL/min,
   * Serum albumin ≥2.5 g/dL,
   * Total bilirubin ≤1.5 × ULN (<3 ULN if Gilbert's disease),
   * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN. If the participant has liver metastases, ALT and AST < 5 × ULN, he/she will be eligible for the study,
   * Adequate blood clotting function: defined as an international normalized ratio/prothrombin time ≤1.5 × ULN and either partial thromboplastin time or activated partial thromboplastin time within normal limits.

   Note: Transfusion (red blood cell or platelet) or G-CSF administration is not allowed within 14 days prior to the day on which bone marrow function is assessed, or at any time after this day and prior to cycle 1 day 1.
7. Women of childbearing potential must have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) result within 3 days of enrolment.
8. Men or women of childbearing potential must agree to the use of effective contraceptive for the study duration and for at least 7 months after the last dose of study treatment for women, and at least 4 months for men.
9. Patient must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion criteria:

1. AI resistant patients who are eligible to SAFIR 03 - ARRIBA trial (i.e. PIK3CA mutated patients), until SAFIR 03 - ARRIBA study closure or study steering committee's decision.
2. Patient has received more than 2 cycles of the ongoing CDK4/6 inhibitor treatment combined with either AI or fulvestrant.
3. Patient has interrupted the ongoing CDK4/6 inhibitor treatment for more than 14 days.
4. Patient has evidence of clinical or radiological disease progression.
5. Patient has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline.

   Note: Patients may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to enrolment and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as: Chemotherapy-induced neuropathy and fatigue.
6. Patient has malignancies within 3 years, other than that under study, with the exception of: adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.
7. Patient is at high medical risk because of severe or uncontrolled systemic disease, such as uncontrolled diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, chronic pancreatitis, chronic active infection with hepatitis B virus, hepatitis C virus, or HIV, active untreated or uncontrolled fungal, bacterial or viral infections, active primary immunodeficiency etc.
8. Uncontrolled or significant cardiovascular disease, including any of the following:

   * History of myocardial infarction within 6 months before enrolment,
   * History of symptomatic congestive heart failure (New York Heart Association Class II to IV),
   * Patient with a corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (males) based on average of the screening triplicate12-lead ECG,
   * Patients with known troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrolment to rule out myocardial infarction.
9. Clinically severe pulmonary compromise resulting from current pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months of the study enrolment, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (i.e., rheumatoid arthritis, Sjögren's, sarcoidosis, etc.), or prior pneumonectomy.
10. Patient has spinal cord compression or clinically active central nervous system metastases, defined as untreated or symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
11. Major surgery within 4 weeks before study enrolment.
12. Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to enrolment, or who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow was irradiated
13. Patient using drugs that could have pharmacokinetics interaction with investigational drugs. Concomitant use of strong CYP3A4 inhibitors or OATP 1B inhibitors should be avoided. If concomitant use of strong CYP3A4 or OATP 1B inhibitors is unavoidable, consider delaying T-DXd treatment until the inhibitors have cleared from the circulation (approximately 3 elimination half-lives of the inhibitors) when possible. If a strong CYP3A4 inhibitor or an OATP 1B inhibitor is co-administered and T-DXd treatment cannot be delayed, patients should be closely monitored for adverse reactions.
14. Patient receiving drug that may cause QTc prolongations or cardiac arrhythmia. Pimozide (Orap®) and cisapride (Prepulsid®) are strictly contraindicated: they are associated with a major risk of ventricular rhythm disorder.
15. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of T-DXd.
16. Participation in a therapeutic clinical study within 4 weeks before enrolment.
17. Patient is currently pregnant, breastfeeding, or planning to become pregnant
18. Patient has substance abuse history or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the patient's participation in the clinical study or evaluation of the clinical study results.
19. Person deprived of their liberty or under protective custody or guardianship.
20. Social, familial, or geographic factors that would interfere with study participation or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From first treatment administration to disease progression or death, up to 5 years
  The progression-free survival is the length of time during and after treatment of the disease with T-DXd that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival (OS) | From the first T-DXd administration to death due to any cause, up to 5 years
  The overall survival is the length of time from first T-DXd administration that patients enrolled in the study are still alive.
Objective response Rate (ORR) | From first T-DXd Administration to 6 months after the first administration of treatment, up to 5 years
  The objective response rate is defined as the percentage of patients with a complete response (CR) or a partial response (PR) for a T-DXd treatment.
Duration of response (DoR) | From the date of first documentation to disease progression or death, up to 5 years
  The time from first documented response (CR or PR) until the date of the first disease progression or death from any cause, whichever occurs first.
Clinical benefit rate (CBR) | From first T-DXd Administration to 6 months after the first administration of treatment, up to 5 years
  The clinical benefit risk is defined as the proportion of patients with at least a confirmed CR, PR, or a stable disease for 6 months or more after the first administration of treatment.
Time to response (TTR) | From the first T-DXd administration to objective response, up to 5 years
  The time to response is defined as the time from the first T-DXd administration to the first documentation of CR or PR.
Toxicity during the study | Throughout study completion, up to 5 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice ANDRE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (34):
- France (34):
  - Chu Amiens Picardie, Amiens
  - Clinique de L'Europe Amiens - Cthe, Amiens
  - Centre Hospitalier D'Auxerre, Auxerre
  - Sainte Catherine Institut Du Cancer Avignon Provence, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - Hôpital Simone Veil de Blois, Blois
  - Chu de Brest - Hôpital Cavale Blanche, Brest
  - Clinique Pasteur Lanroze - Cfro - Groupe Vivalto Sante, Brest
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier de Cholet, Cholet
  - Pôle Santé République (Elsan), Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Chi Fréjus-Saint-Raphaël, Fréjus
  - Chd Vendée, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Clinique de La Sauvegarde, Lyon
  - Institut Paoli Calmettes, Marseille
  - Icm Val D'Aurelle, Montpellier
  - Medipôle de Nancy - Cog-Ilc (Polyclinique de Gentilly), Nancy
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Centre Hospitalier de Pau, Pau
  - Hopital Privé Des Côtes D'Armor (Hpca) - Cario, Plérin
  - Institut Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Chp Saint-Grégoire - Groupe Vivalto Sante, Saint-Grégoire
  - Clinique Sainte-Anne - Gh Saint-Vincent, Strasbourg
  - Hôpitaux Du Léman, Thonon-les-Bains
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No